CLINICAL TRIAL: NCT05156580
Title: Long-term Impact of Overweight/Obesity and Hypertension on Cardiovascular Risk in Middle-aged and Elderly Adults: A Cohort Study
Brief Title: Tongzhou Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Tongzhou Yongshun Community Health Service (Unknown); Beijing Tongzhou Lucheng Community Health Service (Unknown); Beijing Tongzhou Xuxinzhuang Community Health Service (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-P2-163-01
Record Dates: First submitted 2021-11-24; First posted 2021-12-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Hypertension
Keywords: Obesity; Hypertension; Cardiovascular risk
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Obese hypertensive group: Patients who were diagnosed with obesity (body mass index (BMI)≥28kg/m2) and hypertension (systolic blood pressure (SBP)/diastolic blood pressure (DBP) ≥ 140/90 mmHg).
  Interventions: Other: No intervention
- Overweight hypertensive group: Overweight patients (24 kg/m2≤BMI≤28 kg/m2) diagnosed with hypertension (SBP/DBP≥140/90 mmHg).
  Interventions: Other: No intervention
- Lean hypertensive group: Lean patients (BMI ≤ 24 kg/m2) diagnosed with hypertension (SBP/DBP ≥ 140/90 mmHg).
  Interventions: Other: No intervention
- Lean normotensive: Lean patients (BMI ≤ 24 kg/m2) diagnosed with normotensive (SBP/DBP < 140/90 mmHg).
  Interventions: Other: No intervention
- Overweight normotensive: Overweight patients (24 kg/m2≤BMI≤28 kg/m2) diagnosed with normotensive (SBP/DBP<140/90 mmHg)
  Interventions: Other: No intervention
- Obese normotensive: Patients who were diagnosed with obesity (BMI≥28kg/m2) and normotensive (SBP/DBP<140/90 mmHg).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study without any intervention

SUMMARY:
Long-term Impact of Overweight/Obesity and Hypertension on Cardiovascular Risk in Middle-aged and Elderly Adults

DETAILED DESCRIPTION:
Overweight and obesity are major risk factors associated with the development of hypertension, poor blood pressure control, and adverse cardiovascular outcomes. However, evidence regarding the long-term impact of overweight/obesity and hypertension on cardiovascular risk in middle-aged and elderly populations remains limited. Therefore, the present study aims to evaluate the long-term effects of overweight/obesity and hypertension on cardiovascular risk in middle-aged and elderly adults.Additionally, a subgroup analysis will be conducted in participants with sarcopenia to assess the influence of blood pressure on prognosis, exploring potential interactions between muscle loss, hypertension, and cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ages of ≥ 45 years
* Participants from routine health examinations at Tongzhou Community Health Service Center
* Availability for follow-up until 2026
* No major barriers to provide written consent

Exclusion Criteria:

* NA

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults undergoing routine physical examinations at community health service centers in Tongzhou, China.
Sampling Method: Non-Probability Sample
Enrollment: 31080 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with major adverse cardiovascular events (MACEs) | 2021-2026
  Percentage of participants with major adverse cardiovascular events (MACEs), including all-cause death, nonfatal myocardial infarction (MI), nonfatal stroke and coronary revascularization.

SECONDARY OUTCOMES:
Percentage of participants with all-cause death | 2021-2026
  Percentage of participants with cardiovascular, non-cardiovascular and undetermined death.
Percentage of participants with MI | 2021-2026
  Percentage of participants with fatal and nonfatal MI.
Percentage of participants with stroke | 2021-2026
  Percentage of participants with fatal and nonfatal stroke.
Percentage of participants undergoing coronary revascularization | 2021-2026
  Percentage of participants undergoing ischemia- and non-ischemia-driven coronary revascularization.
Change in BP control rate | 2021-2026
  Change in BP control rate (office BP: SBP < 140 mmHg and DBP < 90 mmHg) from baseline to follow-up.
Change in SBP | 2021-2026
  Change in SBP from baseline to follow-up.
Change in estimated glomerular filtration rate (eGFR) | 2021-2026
  Change in estimated glomerular filtration rate (eGFR) in ml/min/1.73m2 from baseline to follow-up.
Change in low-density lipoprotein-cholesterol (LDL-c) | 2021-2026
  Change in low-density lipoprotein-cholesterol (LDL-c) in mmol/L from baseline to follow-up.
Percentage of participants with Metabolic dysfunction-associated steatotic liver disease (MASLD) | 2021-2026
  Percentage of participants with Metabolic dysfunction-associated steatotic liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchong Huang, M.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No